CLINICAL TRIAL: NCT02487836
Title: Phase II Trial Evaluating the Efficacy of Laying a Biliary Stent for Producing a Heavy Chemotherapy in Unresectable Pancreatic Adenocarcinomas
Brief Title: Trial Evaluating the Efficacy of Laying a Biliary Stent for Producing a Heavy Chemotherapy in Unresectable Pancreatic Adenocarcinomas
Acronym: PROPAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROPAC-IPC 2012 006
Record Dates: First submitted 2015-06-25; First posted 2015-07-02 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2013-10

CONDITIONS: Adenocarcinoma of Head of Pancreas
Keywords: Laying of the biliary stent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- First attempt stenting (T0 = date of the first act) (Other): Efficacy of laying of a biliary stent for chemotherapy realization
  Interventions: Device: Type WallFlex or Evolution biliary, stent system

INTERVENTIONS:
Device: Type WallFlex or Evolution biliary, stent system — Laying of a stent biliary

SUMMARY:
For many years, the treatment of jaundice due to head pancreatic adenocarcinoma is based on the endoscopic biliary stent. This technique has been shown to be preferable to a surgical shunt.

Recently, adjuvant chemotherapy with FOLFIRINOX regimen (clinical trial) has revolutionized the treatment of metastatic pancreatic adenocarcinoma increasing overall survival in a major way. This design will also be developed in patients with neoadjuvant tumor called "borderline" (the limit of the resectability).

However, several conditions (protocol) are required to consider the implementation of this design : age ≤ 75 years, PS 0 or 1, good hematological parameters and bilirubin ≤ 1.5 times the ULN.

In addition, a randomized study showed that preoperative biliary stent treatment, despite a success rate of 94%, is associated with more complications than surgery fast (related gesture bladder).

It would be interesting to analyze, prospectively, the fate of a series of patients with cancer of the pancreatic head with compression of the lower part of the bile duct, PS 0 or 1 and for which the only limit to FOLFIRINOX design is jaundice or high risk of jaundice.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged > 18 ans and ≤ 75 ans
* Suspicion of adenocarcinoma of the head of the pancreas leading to the placement of a biliary stent
* Either metastatic or "borderline" (at the limit of resectability) or locally advanced
* PS = 0 or 1
* Hematological laboratory parameters (ANC ≥ 1.5 ** 10 9 / l (/ mm3), platelets ≥ 100 ** 10 9 / l (G / L)) and kidney (calculated creatinin clearance> 60 ml / min)
* Jaundice (bilirubin> 20 mmol / L) by compressing the lower part of the bile duct (dilatation of the extrahepatic bile duct)
* Written informed Consent
* Affiliation to social security

Exclusion Criteria:

* Pregnant or lactating woman or without contraception (for child bearing potential women)
* Patient deprived of liberty or under supervision of a guardian
* Impossibility to undergo medical examinations of the study for geographical, social or psychological reasons
* Contra-indication for study procedure
* Predictable technical impossibility to position a stent endoscopically (prior upper GI surgery)
* Life expectancy assumed less than 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Determine the percentage of patients who, at Day 28 after the first attempt stenting (T0 = date of the first act), has received or is able to receive FOLFIRINOX. | At day 28 after the laying of the biliary stent

SECONDARY OUTCOMES:
Rate of biliary infection starting within 3 months after insertion of the prosthesis | From the laying of the biliary stent to 3 months follow up
Prosthetic dysfunction within 3 months (recurrence of jaundice with dilated bile ducts) | From the laying of the biliary stent to 3 months follow up
Complication (s) other (s) (bleeding, perforation, ...) possibly attached (s) endoscopic treatment within 3 months. | From the laying of the biliary stent to 3 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc RAOUL, MD, PHD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, France

REFERENCES:
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr